CLINICAL TRIAL: NCT07159516
Title: Identifying Birth-Related PTSD: Cutoffs for the City Birth Trauma Scale
Status: Completed | Type: Observational
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Hanna Grundström, Principal Investigator, Associate Professor, Region Östergötland
Other Study IDs: Dnr 2023-04534-01
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Childbirth-related PTSD; PTSD; PTSD (Childbirth-Related); PTSD - Post Traumatic Stress Disorder; Post Traumatic Stress
Keywords: PTSD; childbirth; cut-off; CityBits; sensitivity; specificity; Diagnostic Interview; ROC curve
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Individuals recruited from birth units and social media who recently gave birth
  Interventions: Diagnostic Test: Diagnostic interview

INTERVENTIONS:
Diagnostic Test: Diagnostic interview — SCID-5 Clinician Version (SCID-5-CV) was used as gold standard method for determining if diagnostic criteria of PTSD was met or not (First, 2023). SCID-5-CV has been validated for use via telephone with good results for PTSD (Osorio et al., 2019). Only the PTSD-chapter was used, and exclusively birth-related traumatic experiences were considered. This was done achieved by adding a question to the interview guide, addressing potentially traumatic experiences associated with healthcare during a physical examination, operation, intensive care or childbirth.

SUMMARY:
A total of 67 people were recruited from maternity units and social media to take part in the study. They first completed an online questionnaire, then filled out the CityBiTS measure, and finally took part in a diagnostic interview over the phone. The CityBiTS scores were compared to the results of the interviews using ROC curve analysis. We looked at how well the scores identified cases (sensitivity), correctly identified non-cases (specificity), and overall accuracy to find the best cutoff scores and see how these compared to other available methods.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or more
* who had given birth with a minimum at four weeks prior to completing CityBiTS,
* who had a sufficient level of Swedish to participate.

Exclusion Criteria:

* Cases of stillbirth

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Recruitment was performed from a risk group of individuals with a higher likelihood of having BR-PTSD than the average population, to decrease the number of needed diagnostic interviews. Recruitment was made achieved via two different paths. Since birth complications are important risk factors for BR-PTSD, individuals with documented medical complications during birth were recruited from nine birth units in different parts of Sweden for the first path. These were identified by the following diagnostic codes in medical records. Those meeting inclusion criteria were invited by postal mail, including information about the study as well as a link and QR-code to the first survey. The second recruitment path was via social media. The ad invited those who had recently given birth and experienced the birth as difficult.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Number of participants fulfilling the diagnostic criteria for BR-PTSD based on the diagnostic interview compared to CityBiTS | Day 1

SECONDARY OUTCOMES:
Cut-offs for CityBits | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vrinnevisjukhuset, KK, Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: No